CLINICAL TRIAL: NCT00609661
Title: Comparison of Burn Severity and Patient Outcomes to the Subsets of Mesenchymal Stem Cells Identified in the Blood of Burn Victims
Brief Title: Adult Stem Cell Response to Burn Injury
Status: Withdrawn | Type: Observational
Why Stopped: Assay for stem cell analysis not available
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Chandan K Sen, Principal Investigator, Ohio State University
Other Study IDs: 2006H00286
Record Dates: First submitted 2008-01-24; First posted 2008-02-07 (Estimated); Last update posted 2012-10-08 (Estimated); Status verified 2012-10

CONDITIONS: Wound Healing; Burn
Keywords: Mesenchymal Stem Cells, Burn
MeSH Terms: conditions — Burns

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole Blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Patients presenting to the Ohio State University Emergency Department or directly admitted to the Ohio State University Burn Unit following thermal burn.
- 2: Healthy volunteers

SUMMARY:
This study is designed to determine the response of adult stems cells, also referred to as mesenchymal stem cells (MSCs), to tissue injury resulting from thermal burns. The study will consist of a one time collection of a patient's blood, about one teaspoon, on the third day following the initial burn. MSCs in the blood will then be quantitated and identified using according to unique proteins found on their cell surface using flow cytometry. The results of flow cytometry analysis will then be compared to the patients characteristics (age, sex, race, etc.), their past medical history (hx of diabetes, hypertension, heart disease, etc.) and to the patient outcome (length of hospital stay, mortality, etc.).

DETAILED DESCRIPTION:
Traumatic and non-traumatic disease processes result in varying tissue injury that can culminate in organ failure and death. Current literature has demonstrated that adult stem cells (ASCs) are mobilized into peripheral circulation as a heterogeneous population of cells following tissue injury. The significance of this heterogeneity has not yet been defined. Other studies have shown ASCs augment tissue repair under appropriate conditions. This proposal will begin to elucidate the mechanism of ASC activation, mobilization and localization to sites of injury. This study will use flow cytometry to identify subsets of ASCs mobilized in response to tissue injury and compare this response to the patient's demographics, comorbidities, in hospital morbidities, and mortality. Patients with thermal burns will be used as a model of tissue injury given the quantity of tissue injured and the robust signal generated from this injury. ASCs are currently being investigated as adjuncts to tissue repair involving a host of tissues, including cardiac, neural, and renal. The identification of a specific subset of ASCs selectively mobilized in response to tissue injury would alter all studies involving ASCs in tissue repair and necessitate the identification and targeting of subsets selectively mobilized in response to injury to each particular tissue.

ELIGIBILITY:
Inclusion Criteria:

* Any consentable patient presenting to the Ohio State University Emergency Department or directly admitted to the Ohio State University Burn Unit within three days of a thermal burn

Exclusion Criteria:

* Prisoners
* Pregnant patients and nonconsentable patients.

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Any patient who is consented following presentation to the Ohio State University Emergency Department or directly admitted to the Ohio State University Burn Unit within three days of a thermal burn
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2008-02; Primary Completion 2010-02 (Estimated); Study Completion 2010-06 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Chandan K Sen, PhD, Principal Investigator — Ohio State University; Daniel P Zelinski, MD, PhD, Study Director — Ohio State University; Sorabh Khandelwal, MD, Study Director — Ohio State University